CLINICAL TRIAL: NCT00494988
Title: Self-control Trial to Evaluate the Remission Rate and Safety in Newly Diagnosed Type 2 Diabetes Patients After Short-term Intensive Insulin Aspart and Insulin NPH Treatment
Brief Title: Self-control Trial to Evaluate the Remission Rate in Newly Diagnosed Type 2 Diabetes Patients After Treatment With Insulin Aspart
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANA-1635
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin aspart
Drug: insulin NPH

SUMMARY:
This trial is conducted in Asia. The aim of this trial is evaluate the remission rate in newly diagnosed subjects with type 2 diabetes after short-term intensive treatment with insulin aspart and insulin NPH.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes newly diagnosed within 6-12 months
* FBG: 11.1-17.0 mmol/L
* Body mass index (BMI) larger than 25.0 kg/m2

Exclusion Criteria:

* Known or suspected allergy to trial product(s) or related products
* Recurrent major hypoglycaemia as judged by the Investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2004-12; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Remission rate | after 24 weeks

SECONDARY OUTCOMES:
blood glucose profiles
HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Beijing, China

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com